CLINICAL TRIAL: NCT00207623
Title: Evaluation of the Arthritis Basics for Change (ABCs) Self Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: St. Louis University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCCDPHP-SIP 3-01; U88/CCU715766-SIP 3-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis
Keywords: arthritis; self management; patient education
MeSH Terms: conditions — Arthritis

INTERVENTIONS:
Behavioral: Arthritis Basics for Change Education program

SUMMARY:
While there are a variety of arthritis education materials available, the evidence-base on most of them is slim, so it i impossible to know what benefits they may have for the people who participate. The purpose of this project is to evaluate the effectiveness of the mail-delivered self-management education program, Arthritis Basics for Change (ABCS) with an emphasis on changes in knowledge, beliefs, behavior, self efficacy and health outcomes, and to evaluate the appropriateness, usefulness, and readibility of the program. This project will assist CDC's Arthritis Program in determining the usefulness of the ABCs program for helping people with arthritis improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

adults with arthritis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-07; Study Completion 2003-07

PRIMARY OUTCOMES:
Arthritis management knowledge at 6 months
self management beliefs at 6 months
Self management behaviors at 6 months
Self efficacy for arthritis management at 6 months
Health status at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anjali D Despande, PhD, MPH, Principal Investigator — St. Louis University